CLINICAL TRIAL: NCT01151189
Title: A Phase II, Proof of Concept, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Protective Efficacy Against TB Disease, Safety, and Immunogenicity of MVA85A/AERAS-485 in Healthy, HIV-infected Adults
Brief Title: Efficacy Against TB Disease, Safety, and Immunogenicity of MVA85A/AERAS-485 in HIV-Infected Adults (C-030-485)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: University of Oxford (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-030-485
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Tuberculosis; HIV Infections
Keywords: HIV; Tuberculosis; Vaccine
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — MVA 85A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo is a licensed product manufactured by Allermed, Inc. and is used for evaluation of delayed-type of hypersensitivity reactions in adults.
  Interventions: Biological: Placebo
- MVA85A/AERAS-485 (Experimental): MVA85A/AERAS-485 is a recombinant modified vaccinia virus Ankara expressing the M. tuberculosis antigen, Ag85A. Dosage of the study vaccine to be administered will be 1x10^8 pfu.
  Interventions: Biological: MVA85A/AERAS-485

INTERVENTIONS:
Biological: MVA85A/AERAS-485 — Subjects received intradermal injection of MVA85A/AERAS-485 on Study Day 0, followed 6-9 months later by a booster injection of MVA85A/AERAS-485.
  Arms: MVA85A/AERAS-485
Biological: Placebo — Subjects received an intradermal injection placebo on Study Day 0, followed 6-9 months later by a booster injection of placebo.
  Other Names: Candida albicans Skin Test Antigen; Candin
  Arms: Placebo

SUMMARY:
This is a phase II, proof of concept, randomized, double-blind, placebo-controlled study to evaluate the protective efficacy against TB disease, safety, and immunogenicity of MVA85A/AERAS-485 in healthy, HIV-infected adults.

This study consists of 650 adults subjects (ages 18-50 years of age inclusive) who will receive study vaccine or placebo at Study Day 0 and again 6-9 months later. Samples for real-time evaluation of immunogenicity were to be collected from 70 subjects (immunogenicity analysis set).

DETAILED DESCRIPTION:
This Phase II multi-country trial was conducted as a randomized, double-blind, placebo-controlled trial in 650 HIV-positive adults with no evidence of active TB disease. Subjects were stratified at the time of randomization by whether or not they were receiving anti-retroviral therapy (ART) and then randomized in a ratio of 1:1 to receive either MVA85A/AERAS-485 at 1 x 10^8 plaque forming units (pfu) or placebo (Candin). Randomization of each group was capped so that at least 50% of the subjects randomized were receiving ART at randomization. Subjects were to receive an intradermal injection of MVA85A/AERAS-485 or placebo on Study Day 0, followed 6-9 months later by a booster injection of MVA85A/AERAS-485 or placebo. The minimum follow-up period for each subject was 6 months after their last vaccination, during which subjects were followed for safety, clinical signs and symptoms of TB, and immunogenicity. All subjects were to continue to be followed every 3 months until the last subject enrolled had been followed for 6 months after their last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the written informed consent process prior to undergoing any screening evaluations.
* Either males or females aged 18-50 years (inclusive) on Study Day 0
* In general good health, confirmed by medical history and physical examination
* Has ability to complete follow-up period as required by the protocol
* Has laboratory evidence of human immunodeficiency virus (HIV) infection, defined as a positive HIV-1 ELISA test plus a positive confirmatory test (e.g., a second HIV-1 ELISA, polymerase chain reaction (PCR), or rapid ELISA) diagnosed prior to randomization
* Is willing to allow the investigators to discuss the subject's medical history with the subject's HIV physician
* Has 2 CD4+ lymphocyte count test results >350 cells/mm3, performed at least 4 weeks apart, one performed within 6 months prior to randomization and one within 30 days prior to randomization
* Has either: a) a negative QuantiFERON-TB Gold In-Tube test result and tuberculin purified protein derivative (PPD) skin test ≤5 mm induration within 30 days prior to randomization or; b) a positive QuantiFERON-TB Gold In-Tube test result and/or tuberculin PPD skin test >5 mm and has completed 6 months of isoniazid preventive therapy prior to randomization or; c) a positive QuantiFERON-TB Gold In-Tube test result and/or tuberculin PPD skin test >5 mm and has completed treatment for TB disease within 3 year prior to randomization
* Females: Ability to avoid pregnancy during the trial. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must avoid pregnancy by using an acceptable method of avoiding pregnancy from 28 days prior to administration of the study vaccine through the end of the study. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the use of a condom or a diaphragm combined with spermicide.
* Has completed the written informed consent process for simultaneous enrollment in Aeras Vaccine Development Registry protocol

Exclusion Criteria:

* Acute illness
* Fever (temperature > 37.5°C)
* Significant symptomatic infection
* Any evidence of active tuberculosis (TB) disease, as determined by any clinical, radiological, or microbiology measurements.
* Any AIDS defining illness by WHO criteria
* Has received antiretroviral therapy (ART) in the two months prior to study entry (women who have received ART as part of the Prevention of Mother-to-Child Transmission [PMTCT] program and completed this more than 2 months prior to randomization ARE eligible)
* Use of any investigational or non-registered drug, vaccine or medical device other than the study vaccine within 182 days preceding dosing of study vaccine, or planned use during the study period
* Previous receipt of a recombinant modified vaccinia Ankara (MVA) or fusion protein (FP) vector at any time.
* Is enrolled in any other clinical product trial
* Administration of methotrexate, azathioprine, cyclophosphamide, oral corticosteroids (for corticosteroids, this will mean prednisolone, or equivalent, ≥0.5 mg/kg/day; inhaled and topical steroids are allowed) and other immunosuppressive therapies, or blood products or blood derivatives within the six months prior to randomization
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Presence of any history of cancer [except basal cell carcinoma of the skin and cervical carcinoma in situ], or renal failure
* Evidence of severe depression, schizophrenia or mania
* Pregnant females and females who are breast-feeding
* Any history of anaphylaxis in reaction to vaccination
* Principal investigator assessment of lack of willingness to participate and comply with the protocol, or increase in the participant's risk of adverse outcome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 650 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Souleymane Mboup, Principal Investigator — Hopital Aristide Le Dantec; Robert Wilkinson, Principal Investigator — University of Cape Town; Bernard Landry, Study Director — Aeras
Locations (2):
- Hopital Aristide Le Dantec, Dakar, Senegal
- University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Background] Ndiaye BP, Thienemann F, Ota M, Landry BS, Camara M, Dieye S, Dieye TN, Esmail H, Goliath R, Huygen K, January V, Ndiaye I, Oni T, Raine M, Romano M, Satti I, Sutton S, Thiam A, Wilkinson KA, Mboup S, Wilkinson RJ, McShane H; MVA85A 030 trial investigators. Safety, immunogenicity, and efficacy of the candidate tuberculosis vaccine MVA85A in healthy adults infected with HIV-1: a randomised, placebo-controlled, phase 2 trial. Lancet Respir Med. 2015 Mar;3(3):190-200. doi: 10.1016/S2213-2600(15)00037-5. Epub 2015 Feb 26. PMID 25726088

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The placebo is a licensed product manufactured by Allermed, Inc. and is used for evaluation of delayed-type of hypersensitivity reactions in adults.
  Placebo: Subjects were to receive an intradermal injection placebo on Study Day 0, followed 6-9 months later by a booster injection of placebo.
Period: Overall Study
Arm/Group | Placebo | MVA85A/AERAS-485
Started | 326 | 324
Received Vaccine | 325 | 324
Completed | 311 | 314
Not Completed | 15 | 10

BASELINE CHARACTERISTICS:
Population: Safety:
  All randomized subjects who received a dose of study vaccine, based on actual treatment received.
Groups:
- Placebo: Placebo: Subjects were to receive an intradermal injection placebo on Study Day 0, followed 6-9 months later by a booster injection of placebo.
- Total: Total of all reporting groups
Arm/Group | Placebo | MVA85A/AERAS-485 | Total
Number analyzed (Participants) | 325 | 324 | 649
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (6.61) | 37.7 (6.69) | 37.7 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 265 | 520
  Male | 70 | 59 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 304 | 302 | 606
  Coloured | 21 | 22 | 43
  White | 0 | 0 | 0
  Asian | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Senegal | 179 | 178 | 357
  South Africa | 146 | 146 | 292

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: The primary objective of this study is to evaluate the safety of MVA85A/AERAS-485 compared to placebo in HIV-infected, African adult subjects without active TB disease.
Time Frame: Adverse Events (AEs) are recorded for 28 days post vaccination, Serious Adverse Events (SAEs) for at least 6 months post second vaccination.
Population: Safety:
  All randomized subjects who received a dose of study vaccine, based on actual treatment received.
Measure: Number; unit: percentage of participants with an AE
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 325 | 324
percentage of participants with an AE | 96.0 | 99.1

2. Secondary Outcome: Number of TB Cases
Description: Efficacy of MVA85A/AERAS-485 in the prevention of TB disease compared to control subjects who received placebo in HIV-infected, African adult subjects without active TB disease.
Time Frame: For at least 6 months post second vaccination up to 33 months total follow-up.
Population: Per protocol:
  All randomized subjects who received a dose of study vaccine and had no major protocol deviations, were still ongoing in the study 28 days after Study Day 0, and did not have TB diagnosed within 28 days after Study Day 0.
Measure: Number; unit: participants with TB
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 325 | 320
participants with TB | 9 | 6

3. Secondary Outcome: CD4+ Lymphocyte Counts Before and After Administration of MVA85A/AERAS-485 Compared to Placebo in Anti-retroviral Therapy Negative (ART -)Subjects
Time Frame: Up to 6 months post second vaccination.
Population: Safety:
  All randomized ART negative subjects who received a dose of study vaccine, based on actual treatment received.
Measure: Geometric Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 69 | 67
cells/mm^3
  Baseline | 540.60 (1.333) | 541.10 (1.394)
  Study Visit 8 | 557.39 (1.395) | 484.64 (1.430)

4. Secondary Outcome: CD4+ Lymphocyte Counts Before and After Administration of MVA85A/AERAS-485 Compared to Placebo in ART+ Subjects
Time Frame: Up to 6 months post second vaccination.
Population: Safety:
  All randomized ART positive subjects who received a dose of study vaccine, based on actual treatment received.
Measure: Geometric Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 256 | 257
cells/mm^3
  Baseline | 568.07 (1.387) | 564.27 (1.395)
  Study Visit 8 | 606.07 (1.430) | 604.24 (1.449)

5. Secondary Outcome: HIV-1 Viral Load Before and After Administration of MVA85A/AERAS-485 Compared to Placebo in ART - Participants
Time Frame: Up to 6 months post second vaccination.
Population: Safety:
  All randomized ART - subjects who received a dose of study vaccine, based on actual treatment received.
Measure: Geometric Mean (Standard Deviation); unit: copies/mL
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 68 | 65
copies/mL
  Baseline | 6918.76 (8.673) | 9616.55 (9.783)
  Study Visit 8 | 9090.32 (14.101) | 6437.59 (25.781)

6. Secondary Outcome: HIV-1 Viral Load Before and After Administration of MVA85A/AERAS-485 Compared to Placebo in ART+ Participants.
Time Frame: Up tp 6 months post second vaccination
Population: Safety:
  All randomized ART + subjects who received a dose of study vaccine, based on actual treatment received.
Measure: Geometric Mean (Standard Deviation); unit: copies/mL
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 249 | 253
copies/mL
  Baseline | 26.32 (1.339) | 26.87 (1.500)
  Study visit 8 | 27.30 (1.580) | 29.39 (2.040)

7. Secondary Outcome: Counts of Spot-forming Units After Stimulation With AG85A Peptide Pool.
Description: Immunogenicity of MVA85A/AERAS-485 compared to placebo as described by the ex vivo interferon (IFN)-γ enzyme linked immunospot (ELISpot).
Time Frame: 28 days post second vaccination.
Population: First 70 patients enrolled who also had pre-vaccination results available were analyzed.
Measure: Median (95% Confidence Interval); unit: SFU - background/10^6 PBMC
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 33 | 31
SFU - background/10^6 PBMC | 9.00 [4.00 to 30.00] | 254.00 [92.00 to 462.00]

8. Secondary Outcome: Immunogenicity of MVA85A/AERAS-485 Compared to Placebo as Described by Flow Cytometric Intracellular Cytokine Staining (ICS) of CD4+ and CD8+ T Cells After Stimulation With a Peptide Pool of Mycobacterial Antigens.
Description: The antigen-specific negative control-subtracted response for any cytokine (Interferon gamma [INFγ] , Interleukin 2 [IL2], Interleukin 17 [IL17] and tumor necrosis factor [TNF]).
Time Frame: 7 days post second vaccination.
Population: First 70 patients enrolled who also had pre-vaccination results available were analyzed.
Measure: Median (95% Confidence Interval); unit: Percent responding TCells
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 32 | 31
Percent responding TCells
  CD4+ | 0.14 [0.10 to 0.16] | 0.20 [0.16 to 0.34]
  CD8+ | 0.00 [0.00 to 0.02] | 0.04 [0.01 to 0.04]

9. Secondary Outcome: QuantiFERON (QFN) Conversion Rate in MVA85A/AERAS-485 Recipients Compared to Control Subjects Without a Diagnosis of Tuberculosis During the Trial.
Time Frame: For at least 6 months post second vaccination up to 33 months total follow-up.
Population: Per protocol:
  All randomized subjects who received a dose of study vaccine and had no major protocol deviations, were still ongoing in the study 28 days after Study Day 0, and did not have TB diagnosed within 28 days after Study Day 0 (QFT negative at baseline subgroup).
Measure: Number; unit: participants who converted
Arm/Group | Placebo | MVA85A/AERAS-485
Number analyzed (Participants) | 173 | 186
participants who converted | 40 | 38

ADVERSE EVENTS:
Time Frame: AEs reported 28 after each vaccine. SAEs reported for the duration of the study; for at least 6 months after last vaccine up to 33 months total follow-up.
Arm/Group | Placebo | MVA85A/AERAS-485
Serious Adverse Events (participants affected / at risk) | 17/325 | 17/324
Other Adverse Events (participants affected / at risk) | 310/325 | 320/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=325) | MVA85A/AERAS-485 (N=324)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Eye infection syphilitic (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 2 (3) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Meningorrhagia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/255 (1) | 3/265 (3)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0/255 (0) | 1/265 (1)
Congenital anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Death neonatal (General disorders) | 1/255 (1) | 0/265 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=325) | MVA85A/AERAS-485 (N=324)
Anaemia (Blood and lymphatic system disorders) | 45 (51) | 40 (41)
Leukopenia (Blood and lymphatic system disorders) | 48 (52) | 44 (49)
Neutropenia (Blood and lymphatic system disorders) | 122 (139) | 128 (157)
Headache (Nervous system disorders) | 91 (136) | 121 (177)
Tachycardia (Cardiac disorders) | 15 (16) | 20 (21)
Diastolic hypertension (Vascular disorders) | 51 (61) | 56 (65)
Systolic hypertension (Vascular disorders) | 30 (40) | 45 (51)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 52 (58) | 49 (57)
Nausea (Gastrointestinal disorders) | 37 (45) | 37 (43)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (70) | 85 (111)
Myalgia (Musculoskeletal and connective tissue disorders) | 68 (89) | 127 (174)
Fatigue (General disorders) | 70 (94) | 118 (146)
Injection site discharge (General disorders) | 1 (1) | 22 (23)
Injection site erythema (General disorders) | 8 (8) | 42 (46)
Injection site exfoliation (General disorders) | 111 (145) | 243 (364)
Injection site pain (General disorders) | 95 (128) | 229 (370)
Injection site pruritus (General disorders) | 161 (247) | 243 (420)
Injection site swelling (General disorders) | 11 (13) | 59 (74)
Injection site ulcer (General disorders) | 6 (6) | 106 (130)
Injection site vesicles (General disorders) | 0 (0) | 22 (22)
Injection site warmth (General disorders) | 108 (145) | 180 (271)
Malaise (General disorders) | 59 (77) | 115 (143)
Alanine aminotransferase increased (Investigations) | 39 (41) | 36 (39)
Aspartate aminotransferase increased (Investigations) | 34 (37) | 32 (33)
Blood alkaline phosphatase increased (Investigations) | 39 (40) | 33 (38)
Gamma-glutamyltransferase increased (Investigations) | 46 (48) | 48 (53)
Haemoglobin decreased (Investigations) | 28 (31) | 24 (24)
Neutrophil count decreased (Investigations) | 22 (25) | 31 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No